CLINICAL TRIAL: NCT05862129
Title: Association of Intestinal Microbiota and the Onset of Perianal Abscess Based on 16S RDNA Amplicon Sequencing
Status: Completed | Type: Observational
Sponsor: Xi'an Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2022SF-369
Record Dates: First submitted 2023-05-07; First posted 2023-05-17 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Perianal Abscess

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- observation group: This group will collect rectal secretions and stool samples and pus samples from patients with perianal abscess before treatment, and collect rectal secretions and stool samples from patients again 2 months after treatment according to the diagnosis and treatment guidelines.
  Interventions: Procedure: surgical operation
- control group: This group collected rectal secretions and stool specimens from a healthy population.

INTERVENTIONS:
Procedure: surgical operation — Radical operation for the perianal abscess
  Groups: observation group

SUMMARY:
The goal of this observational study is tolearn the association of gut microflora with the onset of perianal abscesses. The main questions it aims to answer are:

Question 1: To understand the structure of rectal microbial community composition and its relationship with pathogenic bacteria in patients with perianal abscess.

Question 2: Understand the structure of rectal microbial community composition in healthy people.

Participants will be collected with rectal secretions and stool specimens.In addition, patients with perianal abscess should also collect pus samples.

ELIGIBILITY:
Inclusion Criteria:

* Observation group: ① Age between 18-60 years, local resident of Xi'an; ② met the diagnostic criteria for perianal abscess and underwent surgical treatment in our hospital; ③ did not use antibiotics before treatment; ④ himself and his family members were willing to participate in this study and signed informed consent.

Control group: ① Age between 18-60 years, permanent residents in Xi'an; ② had no serious chronic disease, no abnormality in physical examination in the last 1 week; ③ did not use drugs that may affect intestinal flora in the last one month; ④ himself and his family members are willing to participate in the study and sign the informed consent.

Exclusion Criteria:

* Failing to retain the specimens as required

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers who did not keep the specimens as required
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Observation group: the structure and changes of rectal flora before and after treatment | Two months
  Analysis of the intestinal microflora based on 16S rDNA amplicon sequencing
Control group: the structure and changes of rectal flora in healthy population | Two months
  Analysis of the intestinal microflora based on 16S rDNA amplicon sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Xi'an Hospital of Traditional Chinese Medicine, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No